CLINICAL TRIAL: NCT06851377
Title: Expanding NGS Data with Optical Genome Mapping (OGM): More Comprehensive Variant Detection in Children with Unexplained Rare Genetic Disorders
Brief Title: Expanding NGS Data with Optical Genome Mapping (OGM)
Acronym: OGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1089
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Neurodevelopmental Disorder (Diagnosis)
Keywords: Optical Genome Mapping, neurodevelopmental disorders, genome sequencing
MeSH Terms: conditions — Neurodevelopmental Disorders; Disease | interventions — Whole Genome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Expanding NGS data with Optical Genome Mapping (OGM) (Experimental): OGM will be used alongside WGS to improve diagnostics in 60 children with severe NDDs lacking a molecular diagnosis after initial CMA and exome analyses.
  Interventions: Genetic: Optical Genome Mapping (OGM) and Whole Genome Sequencing (WGS); Other: Trascriptome analysis

INTERVENTIONS:
Genetic: Optical Genome Mapping (OGM) and Whole Genome Sequencing (WGS) — After identifying causal SVs via OGM, WGS will determine rearrangement breakpoints and examine nearby genes within 100 kb that may have altered expression due to positional effects.
Other: Trascriptome analysis — Following genomic characterization results, transcriptome analysis will be performed on patient-derived lymphoblastoid B-cell lines or fibroblasts to investigate the molecular implications of candidate SVs found in the OGM analysis and identify potential transcriptome abnormalities, such as splicing variants, in patients with atypical clinical features.

SUMMARY:
Over 50% of pediatric neurological and neurodevelopmental disorders lack a molecular diagnosis after standard DNA sequencing and molecular karyotyping. This is due to technical limitations, incomplete variant interpretation, and inadequate genotype-phenotype correlations. New sequencing technologies are crucial for clinical decision-making, offering complete profiles of variants in a patient's DNA to personalize treatment. Optical Genome Mapping (OGM) can detect nearly all structural variants in one experiment. This project aims to use OGM alongside NGS to improve diagnostic yield in 60 children with severe disorders who tested negative for NGS/CMA.

ELIGIBILITY:
Inclusion Criteria:

* individuals without a molecular diagnosis (negative to ES/CMA analyses);
* individuals with genetic diagnoses that explain only one component of their primary phenotype;
* individuals carrying one or more variants of uncertain clinical significance
* individuals with a phenotype highly reminiscent of clinically and molecularly well-defined syndromes (i.e., Marfan Syndrome) but negative to routine molecular analysis.

Exclusion Criteria:

* individuals who have not undergone initial diagnostic genetic tests (ES/CMA)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Genotype-phenotype correlation | once at recruitment
  Number of pathogenic structural variants found by OGM explaining the phenotype

CONTACTS AND LOCATIONS:
Locations (1):
- Cytogenetic Unit of Medical Genetic Laboratory, Bosisio Parini, Lecco, Italy